CLINICAL TRIAL: NCT02860377
Title: Effect of Recorded Maternal Voice on the Emergence of General Anesthesia on Pediatric Patients: a Pilot Study
Brief Title: Maternal Voice on Anesthetic Emergence Period
Acronym: MatherVoice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Eugene Kim, Assistant professor, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DCUMC_1
Record Dates: First submitted 2016-08-03; First posted 2016-08-09 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Anesthesia, General
Keywords: emergence agitation; emergence time; pediatric
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- stranger's voice (Active Comparator): At the end of surgery, patients were stimulated to wake up by recorded stranger's voice, which was recorded before the operation.
  Interventions: Procedure: recorded stranger's voice
- maternal voice (Experimental): At the end of surgery, patients were stimulated to wake up by recorded maternal voice, which was recorded before the operation.
  Interventions: Procedure: recorded maternal voice

INTERVENTIONS:
Procedure: recorded maternal voice — A voice recording will be performed before the operation. At a preoperative visit or preoperative clinic, informed consent was obtained before the recording. On a calm environment, the mother was asked to speak following sentences.
  " OO (first name of child), wake up~. Let's go home with mommy. OO, wake up~. Open your eyes. Take a deep breath. "
  At the end of surgery, the recorded maternal voice was delivered to the child every 15 seconds until he/she wakes up.
  Arms: maternal voice
Procedure: recorded stranger's voice — A voice recording will be performed before the operation. On a calm environment, a blinded female investigator was asked to speak following sentences.
  " OO (first name of child), wake up~. Let's go home with mommy. OO, wake up~. Open your eyes. Take a deep breath. "
  Arms: stranger's voice

SUMMARY:
Mother spend a large amount of time with their children. It is assumed that mother contributes to their neurological development not only with visual stimuli, but also with auditory stimuli. A recent study revealed that prefrontal cortex can be activated in response to the self-name being spoken by the mother than by a stranger. Therefore, investigators suppose that recorded maternal voice can stimulate the pediatric patients and thereby fasten the emergence from general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 2 and 8 years of American Society of Anesthesiologists physical status (ASA PS) I or II who are planned to receive an operation under general anesthesia

Exclusion Criteria:

* ASA PS III or IV
* with developmental delay or neurological diseases associated with symptoms of agitation
* refusal of consent
* with developmental delay
* with allergy or contraindication to use of ketamine (presence of an active upper respiratory tract infection (URI), increased intracranial pressure, open-globe injury, and a psychiatric or seizure disorder)

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Emergence time | During 1 hour after operation
  time from discontinuation of anesthetics to extubation
Incidence of emergence delirium (ED) | During 30 minutes after PACU admission
  The incidence of emergence delirium (ED) was defined as pediatric anesthesia emergence delirium (PAED) score of >12 or Watcha scale over 3.

SECONDARY OUTCOMES:
peak PAED scale | During 30 minutes after PACU admission
  The PAED scale is a validated observational measure of 5 aspects of child behavior (caregiver eye contact, purposeful movement, evidence of awareness of surroundings, restlessness, and inconsolability). Ratings are summed to produce a total score ranging from 0 to 20; greater scores indicate greater severity.
peak Watcha scale | During 30 minutes after PACU admission
  The Watcha scale is a four-point as followings.
  1. calm
  2. crying, but can be consoled
  3. Crying, cannot be consoled
  4. Agitated and thrashing around
eye opening or purposeful movement time | During 1 hour after operation
  time from discontinuation of anesthetics to spontaneous eye opening
BIS over 60 | During 1 hour after operation
  At the end of operation, investigators stop the anesthetics and carefully watch the bispectral index (BIS) monitor. Simultaneously, investigators check the duration of time from discontinuation of anesthetics until the BIS >60.

OTHER OUTCOMES:
peak FLACC score | During 30 minutes after PACU admission
  Face, legs, activity, cry, and consolability (FLACC) score is checked every 10min after PACU admission.
The amount of analgesic/anesthetic consumption at PACU/ward | During 1 hour at PACU
  The amount of analgesics/anesthetic consumption was checked during hospital admission. At PACU, a total PAED score of >12 or a FLACC scale >4, intravenous fentanyl 0.5 mcg/kg was administered as rescue medication and repeated after 10 min if the agitation does not subside.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kim, MD, Study Director — Daegu Catholic University Medical Center
Locations (1):
- Daegu Catholic University Medical Center, Daegu, South Korea